CLINICAL TRIAL: NCT02802358
Title: Evaluation of Health and Social Interventions Aimed to Old People Discharged From Hospital After a Hip or Wrist Fracture Due to a Fall
Status: Completed | Type: Observational
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Responsible Party: Principal Investigator, JOSE M QUINTANA-LOPEZ, MD PhD, Dr., Hospital Galdakao-Usansolo
Other Study IDs: PI08/90417; 2008111016 (Other Grant/Funding Number: Department of Health of the Basque Country)
Record Dates: First submitted 2016-06-08; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Elderly; Wrist Fracture; Hip Fracture
Keywords: Falls; Functionality
MeSH Terms: conditions — Wrist Fractures; Hip Fractures | interventions — Surgical Procedures, Operative; Immobilization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hip fracture: Patients with a hip fracture due to an accidental fall
  Interventions: Procedure: Surgery or non-invasive procedure (reduction of the fracture, immobilization, stabilization)
- Wrist fracture: Patients with a wrist fracture due to an accidental fall
  Interventions: Procedure: Surgery or non-invasive procedure (reduction of the fracture, immobilization, stabilization)

INTERVENTIONS:
Procedure: Surgery or non-invasive procedure (reduction of the fracture, immobilization, stabilization)

SUMMARY:
Objectives: To describe social and health care provided to our older patients who have been admitted in the emergency department (ED) after suffering from a hip or wrist fracture due to a fall. To compare among the different hospitals and town halls, the health and social care that participants received. To compare the functional dependency and health related quality of life (HRQoL) presented by the patients immediately and six months after a fall.

Methodology: Prospective Cohort study. One hundred and fifty patients suffering from each type of fracture (hip or wrist) will be recruited consecutively in the Basque Health System's participant hospitals sub-project. Within 3 sub-projects, more than 3000 cases are expected to be collected. Data will be collected from ED and hospital clinical records and by means of questionnaires to measure functional dependency (Barthel and Lawton indexes) and HRQoL (SF-36) requesting information on status before the fall, immediately and six months later. In addition to this, data referred to care provided to the patients by traumatologist, rehabilitation or primary care provider as well as social services in their homes after the index episode will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Hip or wrist fracture due to an accidental fall.
* Providing informed consent.

Exclusion Criteria:

* Physical or psychological impairments that would prevent patients from properly completing the questionnaires.
* Syncope.
* No acceptance for taking part in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults aged 65 or older with a hip or wrist fracture due to a fall who attended the ED of the participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 1824 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Questionnaires to measure change in the functionality of the elderly | Before and 6 months after the fall

SECONDARY OUTCOMES:
Questionnaire to measure change in the health-related quality of life of the elderly | Before and 6 months after the fall
Questionnaire to measure change in the performance of activities of daily living | Before and 6 months after the fall